CLINICAL TRIAL: NCT01608815
Title: Immunogenicity and Safety of a Single Dose of SP093 Typhoid Vi Polysaccharide Vaccine Given in Japanese Subjects
Brief Title: Study of a Single Dose of SP093 Typhoid Vi Polysaccharide Vaccine in Japanese Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TYP31 (SFY12079); U1111-1124-7699 (Other: WHO)
Record Dates: First submitted 2012-05-28; First posted 2012-05-31 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-04

CONDITIONS: Salmonella Infections; Typhoid Fever; Bacterial Infections
Keywords: Salmonella infections; Typhoid fever; Bacterial infections; Typhoid vaccine
MeSH Terms: conditions — Salmonella Infections; Typhoid Fever; Bacterial Infections | interventions — Vi polysaccharide vaccine, typhoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental): All participants will receive single dose of typhoid Vi polysaccharide vaccine on Day 0.
  Interventions: Biological: Typhoid Vi polysaccharide

INTERVENTIONS:
Biological: Typhoid Vi polysaccharide — 0.5 mL, Intramuscular
  Other Names: Typhim Vi

SUMMARY:
This study is designed to assess the immunogenicity and safety of typhoid Vi polysaccharide vaccine in Japanese participants to support registration of the product in Japan.

Primary Objective:

To describe the seroconversion rate (percentage of subjects with at least a 4-fold increase of their Vi antibody titer) between Day 0 before vaccination and Day 28 after vaccination with typhoid Vi polysaccharide (SP093) vaccine in subjects aged 2 years and above.

Secondary Objectives:

* To describe the safety profile of a single dose of typhoid Vi polysaccharide vaccine up to 28 days after vaccination, in subjects aged 2 years and above.
* To describe the immune response following a single dose of typhoid Vi polysaccharide vaccine in subjects aged 2 years and above.

DETAILED DESCRIPTION:
All participants will receive a single dose of typhoid Vi polysaccharide vaccine on Day 0 and be assessed for immunogenicity on Day 0 before vaccination and on Day 28 post-vaccination. All participants will be monitored for safety for up to 28 days post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 years and above on the day of inclusion
* For subjects ≥ 20 years of age: Informed consent form has been signed and dated by the subjects. For subjects 2 to 19 years of age: Informed consent form has been signed and dated by the parent or other legally representative. Also subjects 7 to 11 years of age will provide oral assent and subjects 12 to 19 years of age will provide written assent form
* Able to attend all scheduled visits/phone call and to comply with all trial procedures
* For a woman of childbearing potential, use of an effective method of contraception from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination.

Exclusion Criteria:

* Any acute and/or serious disease/illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* History of typhoid fever or Salmonella typhi infection, confirmed either clinically, serologically, or microbiologically
* Known systemic hypersensitivity to any of the vaccine components, or history of a life threatening reaction to a vaccine containing the same substances of the study vaccine
* Known or suspected congenital or current/previous acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroids therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the trial inclusion
* Planned participation in another clinical trial during the present trial period
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response
* Receipt of any vaccine within the four weeks preceding the trial vaccination, except for influenza vaccination, which may be received at least two weeks before the study vaccine
* Planned receipt of any vaccine during the trial period
* Clinical or known serological evidence of systemic illness including hepatitis B, hepatitis C and/or Human immunodeficiency virus (HIV) infection
* Ineligible according to the investigator's clinical judgment
* Known pregnancy, or a positive (serum and/or urine) pregnancy test
* Currently breastfeeding a child
* Known thrombocytopenia, contraindicating intramuscular (IM) vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
* Identified as employee of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family member (i.e., immediate, husband, wife and their children, adopted or natural) of the employees or the Investigator
* Previous vaccination against Salmonella typhi disease with either the trial vaccine or another vaccine.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Aventis K. K.
Locations (3):
- Japan (3):
  - Nagoya, Aichi-ken
  - Osaka, Osaka
  - Shinjuku, Tokyo

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 26 May 2012 to 31 August 2012 at 4 clinic centers in Japan.
Pre-assignment Details: A total of 200 participants who met all of the inclusion and none of the exclusion criteria were vaccinated in this study.
Groups:
- Adults (Group 1): Participants ≥18 years of age received a single dose (0.5 mL) of Typhoid Vi Polysaccharide Vaccine
- Adolescents (Group 2): Participants 12 to 17 years of age received a single dose (0.5 mL) of Typhoid Vi Polysaccharide Vaccine
- Children (Group 3): Participants 2 to 11 years of age received a single dose (0.5 mL) of Typhoid Vi Polysaccharide Vaccine
Period: Overall Study
Arm/Group | Adults (Group 1) | Adolescents (Group 2) | Children (Group 3)
Started | 188 | 7 | 5
Completed | 188 | 7 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adults (Group 1) | Adolescents (Group 2) | Children (Group 3) | Total
Number analyzed (Participants) | 188 | 7 | 5 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 7 | 5 | 12
  Between 18 and 65 years | 188 | 0 | 0 | 188
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.2 (11.4) | 15.6 (2.0) | 5.2 (3.8) | 35.7 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 3 | 1 | 76
  Male | 116 | 4 | 4 | 124
Region of Enrollment [Number; unit: Participants]
  Japan | 188 | 7 | 5 | 200

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With At Least a 4-Fold Rise in Vi Antibody Titers Following Vaccination With a Typhoid Vi Polysaccharide Vaccine
Description: Anti Vi antibodies were measured by Enzyme-Linked ImmunoSorbent Assay (ELISA).
Time Frame: Day 0 (pre-vaccination) to Day 28 (post-vaccination)
Population: Vi antibody titers were assessed in the Immunology Analysis Set.
Measure: Number; unit: Participants
Groups:
- Dolescents (Group 2): Participants 12 to 17 years of age received a single dose (0.5 mL) of Typhoid Vi Polysaccharide Vaccine
Arm/Group | Adults (Group 1) | Dolescents (Group 2) | Children (Group 3)
Number analyzed (Participants) | 188 | 7 | 5
Participants | 173 | 6 [0 to 0] | 5 [0 to 0]

2. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies to Vi Antibody Before and Following Vaccination With A Typhoid Vi Polysaccharide Vaccine
Description: Anti-Vi antibodies were measured by enzyme-linked immunosorbent assay (ELISA)
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Geometric Mean Titers were assessed in the Immunology Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Adults (Group 1) | Adolescents (Group 2) | Children (Group 3)
Number analyzed (Participants) | 188 | 7 | 5
Titers
  GMT (pre-vaccination) | 6.6 [5.8 to 7.4] | 10.2 [2.9 to 35.9] | 3.7 [NA to NA] — The 95% Confidence Interval was not calculated as the titer values are less than the Lower Level of Quantitation
  GMT (post-vaccination) | 148.6 [126.9 to 174.0] | 320.0 [230.6 to 444.2] | 501.7 [305.3 to 824.5]

3. Secondary Outcome: Geometric Mean Titer Ratios (GMTRs) of Antibodies to Vi Antibody Following Vaccination With A Typhoid Vi Polysaccharide Vaccine
Description: Anti-Vi antibodies were measured by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 28 post-vaccination
Population: Geometric Mean Titer Ratios were assessed in the Immunology Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Adults (Group 1) | Adolescents (Group 2) | Children (Group 3)
Number analyzed (Participants) | 188 | 7 | 5
Ratio | 22.6 [19.1 to 26.8] | 31.4 [9.2 to 107.9] | 135.6 [82.5 to 222.8]

4. Secondary Outcome: Number of Participants Reporting A Solicited Injection Site or Systemic Reactions Following Vaccination With A Typhoid Vi Polysaccharide Vaccine
Description: Solicited injection site: Pain, Erythema, and Swelling; Solicited systemic reactions: Fever (Temperature), Headache, Malaise, Myalgia. Grade 3 injection site (children): Pain Incapacitating, unable to perform usual activities; Erythema and Swelling ≥ 50 mm; Grade 3 injection site (adults and adolescents): Pain, Significant, prevents daily activity; Erythema and Swelling, >100 mm. Grade 3 systemic reactions: Fever, ≥39˚C; Headache, Malaise, and Myalgia, Significant, prevents daily activity.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Solicited injection site reactions and systemic reactions were assessed in the Safety Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Adults (Group 1) | Adolescents (Group 2) | Children (Group 3)
Number analyzed (Participants) | 188 | 7 | 5
Participants
  Injection site Pain | 139 | 6 [0 to 0] | 3 [0 to 0]
  Grade 3 Injection site Pain | 0 | 0 [0 to 0] | 0 [0 to 0]
  Injection site Erythema | 0 | 0 [0 to 0] | 2 [0 to 0]
  Grade 3 Injection site Erythema | 0 | 0 [0 to 0] | 0 [0 to 0]
  Injection site Swelling | 1 | 0 [0 to 0] | 0 [0 to 0]
  Grade 3 Injection site Swelling | 0 | 0 [0 to 0] | 0 [0 to 0]
  Fever | 2 | 0 [0 to 0] | 1 [0 to 0]
  Grade 3 Fever | 0 | 0 [0 to 0] | 0 [0 to 0]
  Headache | 14 | 0 [0 to 0] | 0 [0 to 0]
  Grade 3 Headache | 1 | 0 [0 to 0] | 0 [0 to 0]
  Malaise | 23 | 0 [0 to 0] | 0 [0 to 0]
  Grade 3 Malaise | 2 | 0 [0 to 0] | 0 [0 to 0]
  Myalgia | 93 | 4 [0 to 0] | 1 [0 to 0]
  Grade 3 Myalgia | 2 | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post vaccination) up to Day 28 post vaccination.
Groups:
- Adults (Group 1): Participants ≥18 years of age received a single dose of Typhoid Vi Polysaccharide Vaccine
- Adolescents (Group 2): Participants 12 to 17 years of age received a single dose of Typhoid Vi Polysaccharide Vaccine
- Children (Group 3): Participants 2 to 11 years of age received a single dose of Typhoid Vi Polysaccharide Vaccine
Arm/Group | Adults (Group 1) | Adolescents (Group 2) | Children (Group 3)
Serious Adverse Events (participants affected / at risk) | 1/188 | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 139/188 | 6/7 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults (Group 1) (N=188) | Adolescents (Group 2) (N=7) | Children (Group 3) (N=5)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults (Group 1) (N=188) | Adolescents (Group 2) (N=7) | Children (Group 3) (N=5)
Nasopharyngitis (Infections and infestations) | 7 (7) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Injection site Pain (General disorders) | 139 (139) | 6 (6) | 3 (3)
Injection site Erythema (General disorders) | 0 (0) | 0 (0) | 2 (2)
Fever (General disorders) | 2 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 14 (14) | 0 (0) | 0 (0)
Malaise (General disorders) | 23 (23) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 93 (93) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.